CLINICAL TRIAL: NCT00086268
Title: Non-small Cell Lung Cancer Study US75 (Z-PACT)
Acronym: ZPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446EUS75; US 75; NCT00093717 (obsolete NCT alias)
Record Dates: First submitted 2004-06-29; First posted 2004-07-01 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: lung cancer; ZPACT; US75; Bone Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Zoledronic Acid; Docetaxel; Carboplatin

ARMS (2):
- Zometa® (Experimental): 4mg monthly for 12 months from date of first chemotherapy dose
  Interventions: Drug: zoledronic acid; Drug: Taxotere; Drug: Carboplatin
- no further treatment (No Intervention): Control arm; no further treatment. Follow-up monthly for 12 months from date of first chemotherapy dose

INTERVENTIONS:
Drug: zoledronic acid
  Arms: Zometa®
Drug: Taxotere
  Arms: Zometa®
Drug: Carboplatin
  Arms: Zometa®

SUMMARY:
This study will evaluate the effects of an investigational drug in combination with chemotherapy in patients with stage IIIB/IV non-small cell lung cancer. This study will measure the effects of this combination on progression of lung cancer, cancer response to treatments, and development of cancer-related bone lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients at least of 18 years old
* Patients with diagnosed non-small cell lung cancer that cannot be treated by surgery
* Women must not be pregnant or attempting to become pregnant
* Able and willing to sign informed consent

Exclusion Criteria:

* Patients with cancer that has spread to the bone
* Patients with cancer that has spread to the brain who are receiving treatment
* Patients with kidney disease
* Patients treated with other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (80):
- United States (80):
  - Clinical Research Consultants, Hoover, Alabama
  - Arizona Oncology Assoc., Tucson, Arizona
  - NEA Clinic, Jonesboro, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - NorthBay Cancer Center, Fairfield, California
  - UCLA, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Med. Oncology Care Associates, Orange, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Cancer Center of Colorado Springs, Colorado Springs, Colorado
  - Northern Hematology-Oncology, Thornton, Colorado
  - Lynn Regional Cancer Center, Boca Raton, Florida
  - New Hope Cancer Centers, Hudson, Florida
  - Oceola Cancer Center, Kissimmee, Florida
  - VA Medical Center, Miami, Florida
  - Innovative Medical Research of South Florida, Inc., Miami Shores, Florida
  - NCH Healthcare System Oncology Research, Naples, Florida
  - Metcare Oncology, Ormond Beach, Florida
  - Hematology-Oncology Associates, Pensacola, Florida
  - AMIT SHAH Medical Group, Sebring, Florida
  - Peachtree Hematology & Oncology, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Straub Clinic & Hospital, Honolulu, Hawaii
  - Kaiser Foundation Hospital, Honolulu, Hawaii
  - Advocate Illinois Masonic Medical Center Creticos Cancer Center, Chicago, Illinois
  - OSF Center for Cancer Care, Rockford, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Community Hospital, Cancer Research Dept., Munster, Indiana
  - Northern Indiana Oncology Associates, South Bend, Indiana
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Kansas City Cancer Ctr. South, Lenexa, Kansas
  - Hematology/Oncology Clinic, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Oncology Care Associates, Bethesda, Maryland
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Kalamazoo Hematology & Oncology, Kalamazoo, Michigan
  - Mitchell Folbe, MD, PC, Troy, Michigan
  - Park Nicollett Institute, Saint Louis Park, Minnesota
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Odyssey Research, Scottsbluff, Nebraska
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - East Orange VA Medical System, East Orange, New Jersey
  - Howell Office Plaza, Howell Township, New Jersey
  - Atlantic Hem Onc Associates, LLC, Manasquan, New Jersey
  - Hematology/Oncology Assoc. of South Jersey, Mount Holly, New Jersey
  - Cancer Institute of New Jersey at Cooper University Hospital, Voorhees Township, New Jersey
  - New Mexico Oncology Hematology Consultants, Ltd., Albuquerque, New Mexico
  - San Juan Regional Cancer Ctr., Farmington, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Engracio Cortes, MD, Bayside, New York
  - Arena Oncology Assoc., Great Neck, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Southern Oncology Research, Grifton, North Carolina
  - Barberton Citizens Hospital-Cancer Center, Barberton, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Forum Health Cancer CareCenter, Youngstown, Ohio
  - Cancer Specialists of Oklahoma, Oklahoma City, Oklahoma
  - Hematology Oncology Associates, Medford, Oregon
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Charleston Cancer Center, Charleston, South Carolina
  - Liberty Hematology-Oncology, Columbia, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Knoxville Cancer Center, Knoxville, Tennessee
  - Cancer Specialists of South Texas, Corpus Christi, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Tyler Hematology Oncology, PA, Tyler, Texas
  - Odyssey Research, Belle Haven, Virginia
  - Masoom Kandahari, MD, Woodbridge, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Result] Pandya KJ, Gajra A, Warsi GM, Argonza-Aviles E, Ericson SG, Wozniak AJ. Multicenter, randomized, phase 2 study of zoledronic acid in combination with docetaxel and carboplatin in patients with unresectable stage IIIB or stage IV non-small cell lung cancer. Lung Cancer. 2010 Mar;67(3):330-8. doi: 10.1016/j.lungcan.2009.04.020. Epub 2009 Jun 2. PMID 19493585